CLINICAL TRIAL: NCT02757586
Title: Resistances of CLL and Treatment of CLL
Brief Title: Treatment of Chronic Lymphocytic Leukemia
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Peking University People's Hospital (Other)
Collaborators: Beijing Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: Study on CLL
Record Dates: First submitted 2016-04-17; First posted 2016-05-02 (Estimated); Last update posted 2016-05-13 (Estimated); Status verified 2016-05

CONDITIONS: Leukemia, Lymphocytic, Chronic, B-Cell
Keywords: chronic lymphocytic leukemia; XPO1; in vitro; in vivo
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — RNA, Small Interfering

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — PB
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Genetic: shRNA — Using shRNA interfered the expression of the gene of CLL

SUMMARY:
CLL is a disease of the elderly, identifying effective therapies with better toxicity profiles is thus a high priority, and targeted therapies may allow attainment of this goal.

DETAILED DESCRIPTION:
Chronic lymphocytic leukemia (CLL) is a common adult leukemia characterized by the extensive accumulation of monoclonal, relatively mature CD5+CD23+ B lymphocytes in lymphoid organs, bone marrow, and peripheral blood. CLL cells accumulate because of defective apoptosis, which extends survival. CLL is a heterogeneous disease. Chemoimmunotherapy is the standard front-line approach for patients younger than 65 years with CLL, with the combination of fludarabine, cyclophosphamide, and rituximab used most commonly. Some CLL patients do not respond well to routine chemoimmunotherapy. Despite recent advances in the treatment of CLL by use of modern chemoimmunotherapy, the disease remains incurable for most patients with the exception of those who have the option of an allogeneic transplantation. However, treatments with chemoimmunotherapy are associated with significant toxicities and sustained immunosuppression, and the rates of myelosuppression and infection are high. Such complications are more frequent and more severe in patients older than 65 years because of reduced marrow reserve, and presence of comorbidities. Because CLL is a disease of the elderly, identifying effective therapies with better toxicity profiles is thus a high priority, and targeted therapies may allow attainment of this goal.

CLL tumor cells are highly dependent on the microenvironment where cytokines (eg, CD40L, BAFF, IL-4, IL-6), and contact (eg, stromal cells) promote cell activation and proliferation, and also resistance to spontaneous and drug-mediated apoptosis. Many of these microenvironment-activated pathways merge with TSPs exported by XPO1. XPO1 is therefore a highly attractive molecular target to explore in CLL, because it impacts multiple antitumor and growth suppressive signaling pathways that are dysregulated in this disease.

The investigators therefore hypothesized that a selective XPO1 inhibitor would show efficacy with an acceptable therapeutic index in CLL and other diseases. Indeed, XPO1 inhibition in normal cells (ie, possessing an intact genome) leads to transient cell cycle arrest without cytotoxicity, followed by fast recovery after the drug is removed. To date, efforts to clinically pharmacologically inhibit XPO1 have been unsuccessful because of off-target effects. A selective XPO1 antagonist may allow targeting of the TSPs axes in tumor cells.

ELIGIBILITY:
Inclusion Criteria:

* patients with CLL

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: CLL patients
Sampling Method: Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2016-12; Primary Completion 2018-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
overall response | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Xiao-Jun Huang, Principal Investigator — professor

IPD SHARING:
Plan to Share IPD: Undecided